CLINICAL TRIAL: NCT04027023
Title: Pilot Study for Evaluation of the Impact of Intensive Short-Term Drug Therapy on Beta-Cell Function and Insulin Resistance in Patients With Type 2 Diabetes Mellitus
Brief Title: Evaluation of the Impact of Intensive Short-Term Drug Therapy in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sciema UG (Other)
Collaborators: Innovative Diabetes Treatment Studies LLC. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCTI-DET-001
Record Dates: First submitted 2019-07-11; First posted 2019-07-19 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: open-label, prospective, phase IV study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Diabetes mellitus Type 2 De-escalation treatment (DET) — All employed drugs are approved in the US for treatment of type 2 diabetes and are used within their label. There will be defined individual treatment drug combinations at an earlier stage of diabetes as in standard treatment. The DET combination will be composed out of one each or more of the drugs and interventions listed below.
  A. Relieve for the insulin-producing ß-cells insulin glargine (6 to 20 U at bedtime) insulin degludec (5 to 15 U at bedtime) B. Reduction of hormonal visceral lipid tissue activity/chronic inflammation Weight loss liraglutide (0.6 mg/day) exenatide (15 µg/day) C. Treatment of metabolic and vascular insulin resistance Pioglitazone (30 mg) D. Treatment of glucose toxicity Empagliflozin (SGLT-II inhibitor; 10 mg) Dapagliflozin (SGLTII-Inhibitor, 10 mg) Canagliflozin (SGLT-II inhibitor, 100 mg) Metformin (inhibition of hepatic glucose production, 500 mg)
  To avoid hypos, all drugs are initially given in the lowest possible dose.

SUMMARY:
This phase IV study is a prospective open-label multi-center study to investigate the effect of a temporary individualized poly-pharmaceutical De-escalation treatment with the target to regenerate ß-cell function over 12 weeks on the disease stage and glycemic control in patients with type 2 diabetes. This is an uncontrolled pilot study to collect data for later confirmatory trials.

DETAILED DESCRIPTION:
During the screening visit the patient will arrive at the study site and written informed consent will be obtained by the investigator. Inclusion and exclusion criteria will be controlled and blood will be drawn for HbA1c, the efficacy and the safety parameters. A POCT pregnancy test will be conducted in women of childbearing age. Patient demographics and history will be collect and a physical examination will be performed. The patient will complete a QoL questionnaire and will receive training about the de-escalation therapy approach. After all necessary biomarker results of the screening visit are accessible for the selection of the De-escalation treatment the treatment initiation visit will be performed. During this visit the investigator will use these results to determine a most optimal personalized treatment combination for regeneration of the pancreatic ß-cells within the next three months. An ECG will be recorded and the patient will be informed about his/her personalized treatment and its execution. The patient will receive the drugs in the volume required until the next visit. During the next two visits the patient will arrive at the investigational site at the agreed time-point and information regarding potential adverse events will be collected. Vital signs will be measured, and blood will be drawn for assessment of the efficacy parameters. Information about hypoglycaemia will be collected, and the patient will receive drug supply that lasts until the next visit. The patient will be instructed to stop the anti-diabetic medication 3 days before the next visit.

For the final visit (visit 5) the patient will arrive at the investigational site after an overnight fast and information regarding potential adverse events and hypoglycaemic events will be collected. Vital signs will be measured, and blood will be drawn for assessment of the efficacy parameters. An oral glucose challenge with 75 g of glucose will be conducted with blood draws for assessment of glucose and other biomarkers at time-points 0, 1h and 2h. The investigator will give a recommendation for the consecutive follow-up treatment requirements based on the results of the glucose challenge test. The patient will complete a QoL questionnaire (DTSQ) and this concludes study participation for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained prior to any trial-related activities
* Male or female > 18 years
* Diagnosed with 2 Diabetes
* HbA1c <10%
* Current treatment with diet and exercise or up to two anti-diabetic drugs

Exclusion Criteria:

* Patients participating in another investigational drug study
* Drug or alcohol abuse
* Pregnancy or breast feeding
* Sexually active woman of childbearing age not practicing accepted birth control
* Severe diabetes complications (in the discretion of investigator)
* Unstable significant cardiovascular disease with admission to emergency room or hospital in last 45 days
* Lack of compliance or other reason that in the discretion of the investigator precludes satisfactory participation in the study
* Any severe illness preventing participation in the study per protocol (in the discretion of the investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
impact of a temporary personalized poly-pharmaceutical treatment on the disease stage in patients with type 2 diabetes | 12 weeks
  combined drug application

SECONDARY OUTCOMES:
HbA1c measurement to evaluate the impact of the poly-pharmaceutical treatment on the glycemic control | 12 weeks
  venous blood draw to evaluate the HbA1c
RBP4 will be measured to evaluate the impact of the poly-pharmaceutical treatment on the RBP4 level | 12 weeks
  blood draw to measure the above mentioned biomarker
the biomarker adiponectin will be measured to evaluate the impact of the poly-pharmaceutical treatment on the adiponectin level | 12 weeks
  blood draw to measure the above mentioned biomarker
insulin, c-peptide, intact proinsulin, glucagon will be measured to evaluate the impact of a temporary personalized poly-pharmaceutical treatment on beta-cell function | 12 weeks
  blood draw to measure the above mentioned biomarkers
hsCRP, IL-6, angiopoetin 2 will be measured to evaluate the impact of a temporary personalized poly-pharmaceutical treatment on biomarkers of inflammation | 12 weeks
  blood draw to measure the above mentioned biomarkers
Questionnaire about the diabetes treatment satisfaction (DTSQ) will be filled by the patient to evaluate the impact of a temporary personalized poly-pharmaceutical treatment on the quality of Life | 12 weeks
  Questionnaire to be filled by study participant, the scale of the questionnaire reaches from 1 (very good) to 10 (very bad), all questions are bloning to the diabetes treatment.
Renal function | 12 weeks
  blood draw and urine sample to measure renal function, which will be evaluated with the following parameters creatinine, GFR, total protein (serum and urine), Uric acid and urea before and after the temporary personalized poly-pharmaceutical treatment
Liver function | 12 weeks
  blood draw to measure Liver function, which will be evaluated with the following parameters AST, ALT, gamma-GT, and alkaline phosphatase before and after the temporary personalized poly-pharmaceutical treatment
Heart function | 12 weeks
  blood draw to measure Heart function, which will be evaluated with the following parameters creatine kinase, and cK-MB before and after the temporary personalized poly-pharmaceutical treatment
Electrolytic balance | 12 weeks
  blood draw to measure Electrolytic balance, which will be evaluated with the following parameters: sodium, potassium and calcium before and after the temporary personalized poly-pharmaceutical treatment

CONTACTS AND LOCATIONS:
Locations (2):
- NYC Research, Inc., New York, New York, United States
- Pfützner Science & Health Institute GmbH, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No